CLINICAL TRIAL: NCT03419156
Title: Effect of a Short Message Service Intervention on Patients With Short Bowel Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study ended after review
Sponsor: St. Louis University (Other)
Collaborators: Epharmix, Inc. (Industry)
Responsible Party: Principal Investigator, Yosef Greenspon, MD, Assistant Professor of Surgery; Pediatric Surgery, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 28143
Record Dates: First submitted 2018-01-26; First posted 2018-02-01 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Short Bowel Syndrome
Keywords: text message; telemedicine
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: All patients with SBS on TPN at Cardinal Glennon will receive text messages inquiring about their symptoms instead of weekly phone calls from a nurse. There will be no randomization. All patients will be sent text-messages from the automated system for 6 months to assess response rates and the amount of time saved by the nurse staff. If the patient does not respond to the text messages or the text message responses suggest that the patient may be presenting with potentially harmful symptoms, the nurse will call the patient to inquire about more information.The text messages are designed to help target calls made by the nursing staff.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Text Message Arm (Experimental): Patients in the Text Message Arm will receive a weekly set of text messages inquiring about the patients' symptoms instead of a weekly phone call from the nurse team (standard of care). Potentially harmful symptoms identified by the automated system will generate an alert that will be sent to the medical team. The alert will be immediately sent via email to the nursing team. The nurse will be able to contact the patient to decide the best further treatment. The nurses will check patient response rates daily. If a patient does not respond to their weekly message, then the patient will be called.
  Interventions: Other: Text Message Arm Intervention

INTERVENTIONS:
Other: Text Message Arm Intervention — Patients in the Text Message Arm will receive a weekly set of text messages inquiring about the patients' symptoms instead of a weekly phone call from the nurse team (standard of care). Potentially harmful symptoms identified by the automated system will generate an alert that will be sent to the medical team. The alert will be immediately sent via email to the nursing team. The nurse will be able to contact the patient to decide the best further treatment. The nurses will check patient response rates daily. If a patient does not respond to their weekly message, then the patient will be called.

SUMMARY:
The investigators will be using a text messaging intervention to identify potentially dangerous and re- admission causing symptoms in patients with Short Bowel Syndrome (SBS) on Total Parenteral Nutrition (TPN). Each consented patient will receive weekly text messages inquiring about potentially harmful symptoms identified by a team of physicians. If the patient screens positive via text message, an alert will be sent to the medical team. All patients with SBS on TPN will receive text messages. The investigators will be monitoring response rates to text messages screening for potentially harmful symptoms and compare the text- message response rate to historical rates of successful calls by nurses.

All patients with SBS on TPN will receive text messages instead of weekly phone calls from a nurse. If the patient does not respond to the text messages or the text message responses suggest that the patient may be presenting with potentially harmful symptoms, the nurse will call the patient to inquire about more information.

DETAILED DESCRIPTION:
Short Bowel Syndrome (SBS) is a condition that results from a host of different conditions, the most common of which is Necrotizing Enterocolitis. Patients who have SBS are often Total Parenteral Nutrition (TPN) dependent. TPN is a carefully formulated intravenous nutrition that is utilized either alone or in conjunction with gastrointestinal feeds in patients who fail to achieve adequate caloric intake enterally. According to the American Society of Parenteral and Enteral Nutrition, 360,000 hospital visits required usage of TPN in 2009. Short and long-term use of TPN is associated with catheter infections, cholestasis, liver failure, refeeding-syndrome, hyperglycemia, bone demineralization, and death (1). Thus careful and comprehensive monitoring of patients on TPN, especially after hospital discharge is essential (1-3). Some hospitals have introduced resource intensive support teams consisting of various health care professionals to manage these costly patients (1).

Using a variety of definitions, the incidence of SBS has been estimated at approximately 0.02 to 0.1 percent among all live births (4, 5), 0.5 to 2.0 percent among neonatal intensive care unit (NICU) admissions (4, 5), and 0.7 percent among very low birthweight infants (6). Approximately 80 percent of pediatric SBS cases develop during the neonatal period.

The average cost of care in the US for a single pediatric patient with SBS is $550,250 +/- $248, 398 for the first year of care alone (7). These costs were attributable to prolonged requirements for intensive care resources, numerous surgical procedures, multiple readmissions, TPN and home care during the first year of diagnosis. Interestingly, Spencer et al. suggested that hospital-based costs steadily declined in subsequent years, but home-care services increased every year for the first 5 y of diagnosis (7). This increasing cost was attributable to increasing complications of TPN, especially infectious complications (something our application will specifically try to identify). The mean total cost of care per child over a 5-y period was US$1,619,851 +/- US$1,028,985 (7).

At Cardinal Glenon, a significant amount of time (about 10 hours per week) is spent by nurses calling these patients. This automated system will allow nurses to spend a portion of these 10 hours performing other activities, significantly reducing the costs attributed to SBS patients. Also, most of the mothers of patients who have SBS are between the ages of 15-30. This generation of millennials often have an aversion to phone calls and prefer texts [8]. Text- messages can be answered at a convenient time for the parent while the parent must be present and available to answer a phone call. Multiple prior text message or application intervention studies have reported high response rates, high satisfaction, and improvement in outcomes (9-12). For example, Devitto et al. reported that the estimated odds of reporting critical care symptoms of application group was 8.9 times that of control and showed slightly higher adherence to the prescribed regimen (OR 1.64, 95% CI [1.01, 2.66]) (9). Martinez et al. reported that 16 patients would have returned to the hospital without photos of surgical sites prompting health care team intervention (12). Our automated texting system may improve response rates from these young parents.

For this project, the investigators will be examining the effect of an Epharmix text messaging intervention on identifying potentially dangerous and re-admission causing symptoms with SBS patients on TPN.

ELIGIBILITY:
Inclusion Criteria:

* Patients under the age of 18
* Patients with a diagnosis of short bowel syndrome and who are treated with total parenteral nutrition
* Patients able to understand English or have a caregiver who understands English.
* Patients must have caregiver who has access to a phone (landline or cell phone)

Exclusion Criteria:

* Patients who do not have access to a phone (landline or cell phone), and patients who are not mentally able to consent to the study.
* Patients who are not treated with total parenteral nutrition.
* Patients who do no have a short bowel syndrome diagnosis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Response rate | 6 months
  The primary outcome for this study will be comparing response rates to automated text messages vs historical weekly nurse call success rates. The investigators will compare these values using a chi-square.

SECONDARY OUTCOMES:
Specificity and Sensitivity | 6 months
  Specificity and sensitivity of the alerts generated by the automated system
Cost savings | 6 months
  Cost saved in terms of nurse time required without automated text message intervention
Clinic visits | 6 months
  Number of clinic visits by SBS patients
Readmissions | 6 months
  30 day readmission of SBS patients
Days spent in the hospital | 6 months
  Number of days spent in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Josef Greenspon, MD, Principal Investigator — St. Louis University
Locations (1):
- Cardinal Glennon Children's Medical Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartl WH, Jauch KW, Parhofer K, Rittler P; Working group for developing the guidelines for parenteral nutrition of The German Association for Nutritional Medicine. Complications and monitoring - Guidelines on Parenteral Nutrition, Chapter 11. Ger Med Sci. 2009 Nov 18;7:Doc17. doi: 10.3205/000076. PMID 20049074
- [Background] Duro D, Kamin D, Duggan C. Overview of pediatric short bowel syndrome. J Pediatr Gastroenterol Nutr. 2008 Aug;47 Suppl 1:S33-6. doi: 10.1097/MPG.0b013e3181819007. PMID 18667916
- [Background] Uko V, Radhakrishnan K, Alkhouri N. Short bowel syndrome in children: current and potential therapies. Paediatr Drugs. 2012 Jun 1;14(3):179-88. doi: 10.2165/11594880-000000000-00000. PMID 22452596
- [Background] Salvia G, Guarino A, Terrin G, Cascioli C, Paludetto R, Indrio F, Lega L, Fanaro S, Stronati M, Corvaglia L, Tagliabue P, De Curtis M; Working Group on Neonatal Gastroenterology of the Italian Society of Pediatric Gastroenterology, Hepatology and Nutrition. Neonatal onset intestinal failure: an Italian Multicenter Study. J Pediatr. 2008 Nov;153(5):674-6, 676.e1-2. doi: 10.1016/j.jpeds.2008.05.017. Epub 2008 Jun 27. PMID 18589446
- [Background] Wales PW, de Silva N, Kim J, Lecce L, To T, Moore A. Neonatal short bowel syndrome: population-based estimates of incidence and mortality rates. J Pediatr Surg. 2004 May;39(5):690-5. doi: 10.1016/j.jpedsurg.2004.01.036. PMID 15137001
- [Background] Cole CR, Hansen NI, Higgins RD, Ziegler TR, Stoll BJ; Eunice Kennedy Shriver NICHD Neonatal Research Network. Very low birth weight preterm infants with surgical short bowel syndrome: incidence, morbidity and mortality, and growth outcomes at 18 to 22 months. Pediatrics. 2008 Sep;122(3):e573-82. doi: 10.1542/peds.2007-3449. PMID 18762491
- [Background] Spencer AU, Kovacevich D, McKinney-Barnett M, Hair D, Canham J, Maksym C, Teitelbaum DH. Pediatric short-bowel syndrome: the cost of comprehensive care. Am J Clin Nutr. 2008 Dec;88(6):1552-9. doi: 10.3945/ajcn.2008.26007. PMID 19064515
- [Background] https://www.forbes.com/sites/larryalton/2017/05/11/how-do-millennials-prefer-to- communicate/#58cc85d16d6f
- [Background] DeVito Dabbs A, Song MK, Myers BA, Li R, Hawkins RP, Pilewski JM, Bermudez CA, Aubrecht J, Begey A, Connolly M, Alrawashdeh M, Dew MA. A Randomized Controlled Trial of a Mobile Health Intervention to Promote Self-Management After Lung Transplantation. Am J Transplant. 2016 Jul;16(7):2172-80. doi: 10.1111/ajt.13701. Epub 2016 Mar 14. PMID 26729617
- [Background] Carrier G, Cotte E, Beyer-Berjot L, Faucheron JL, Joris J, Slim K; Groupe Francophone de Rehabilitation Amelioree apres Chirurgie (GRACE). Post-discharge follow-up using text messaging within an enhanced recovery program after colorectal surgery. J Visc Surg. 2016 Aug;153(4):249-52. doi: 10.1016/j.jviscsurg.2016.05.016. Epub 2016 Aug 8. PMID 27423211
- [Background] Cleeland CS, Wang XS, Shi Q, Mendoza TR, Wright SL, Berry MD, Malveaux D, Shah PK, Gning I, Hofstetter WL, Putnam JB Jr, Vaporciyan AA. Automated symptom alerts reduce postoperative symptom severity after cancer surgery: a randomized controlled clinical trial. J Clin Oncol. 2011 Mar 10;29(8):994-1000. doi: 10.1200/JCO.2010.29.8315. Epub 2011 Jan 31. PMID 21282546
- [Background] Martinez-Ramos C, Cerdan MT, Lopez RS. Mobile phone-based telemedicine system for the home follow-up of patients undergoing ambulatory surgery. Telemed J E Health. 2009 Jul-Aug;15(6):531-7. doi: 10.1089/tmj.2009.0003. PMID 19566396